CLINICAL TRIAL: NCT01459263
Title: Mechanochemical Endovenous Ablation of Great Saphenous Vein Incompetence Using the ClariVeinTM Device: a Prospective Study
Brief Title: Early Outcome of Mechanochemical Endovenous Ablation
Acronym: ClariVein-2
Status: Completed | Type: Observational
Sponsor: Rijnstate Hospital (Other)
Collaborators: St. Antonius Hospital (Other)
Responsible Party: Principal Investigator, Michel Reijnen, MD, PhD, Rijnstate Hospital
Other Study IDs: NL26327.091.09
Record Dates: First submitted 2011-08-08; First posted 2011-10-25 (Estimated); Last update posted 2018-04-26 (Actual); Status verified 2018-04

CONDITIONS: Varicosis
Keywords: GSV; insufficiency; ClariVein device; safety; efficacy; QOL

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- GSV insufficiency: Patients with insufficiency of the greater saphenous vein (GSV) will be included.
  Interventions: Device: ClariVein

INTERVENTIONS:
Device: ClariVein — Using the ClariVein device, the GSV will be occluded.

SUMMARY:
More than 25 percent of the general population suffers from varicose veins, which has a considerable impact on quality of life. Nowadays endovenous treatment modalities for great saphenous incompetence are widely accepted. Mechanochemical endovenous ablation is a new tumescent-less technique, that combines mechanical endothelial damage using a rotating wire with the infusion of a liquid sclerosant. The current study aims at evaluating short and long term outcome after mechanochemical endovenous ablation.

ELIGIBILITY:
Inclusion Criteria:

* Insufficiency of the GSV
* Ultrasound criteria for endovenous treatment have been met:
* Diameter GSV between 3-12 mm
* No thrombus present at the GSV part to be treated
* Signed informed consent
* Patient willing to present at follow-up visits
* Age > 18 jaar

Exclusion Criteria:

* Patient is unable to give informed consent
* Patient unable to present at all follow-up visits
* Other treatment is more suitable for the treatment of the varicose veins than mechano-chemical ablation
* Pregnancy and breast feeding
* Known allergy/ contra indication for sclerotherapy
* Previous ipsilateral surgical treatment of varicose veins
* Deep venous vein thrombosis in medical history
* Anticoagulant therapy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with insufficiency of the greater saphenous vein will be included.
Sampling Method: Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2010-11; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Occlusion rate | 30 days, 1, 2, and 5 years
  The percentage of GSV occluded

SECONDARY OUTCOMES:
Health status | 30 days, 1, 2, and 5 years
  Using the RAND 36-Item Short Form Health Survey (SF-36)the general health status will be evaluated at the mentioned time points.
  The SF-36 is a set of generic, coherent, and easily administered quality-of-life measures.
Disease related quality of life | 30 days, 1, 2, and 5 years
  Using the AVVQ (Aberdeen Varicose Vein questionnaire) the quality of life related to the disease will be evaluated at the mentioned time points.
Pain score during procedure | peri-procedural
  The pain will be scored during procedure using the VAS score.
2-weeks post-procedure pain score | two weeks
  The pain will be scored daily for two weeks after the procedure using the VAS score.
recovery time | two weeks
  The time (in days) after the procedure until patients were able to restart daily activity/daily work
procedural complications | during procedure
  all complications related to the procedure will be evaluated at the mentioned time points.
post-procedural complications | 1 year
  all complications related to the procedure will be evaluated at the mentioned time points.

CONTACTS AND LOCATIONS:
Overall Officials: Michel MJ Reijnen, MD, PhD, Principal Investigator — Rijnstate Hospital; Jean-Paul Vries, de, MD, Phd, Principal Investigator — St. Antonius Hospital
Locations (2):
- Netherlands (2):
  - Rijnstate Hospital, Arnhem, Gelderland
  - St. Antonius Hospital, Nieuwegein

REFERENCES:
- [Result] van Eekeren RR, Boersma D, Elias S, Holewijn S, Werson DA, de Vries JP, Reijnen MM. Endovenous mechanochemical ablation of great saphenous vein incompetence using the ClariVein device: a safety study. J Endovasc Ther. 2011 Jun;18(3):328-34. doi: 10.1583/11-3394.1. PMID 21679070
- [Result] van Eekeren RR, Boersma D, de Vries JP, Reijnen MM. [Endovenous mechanochemical ablation for varicose veins--a new endovenous technique without tumescent anaesthesia]. Ned Tijdschr Geneeskd. 2011;155(33):A3177. Dutch. PMID 21854655
- [Result] van Eekeren RR, Boersma D, Konijn V, de Vries JP, Reijnen MM. Postoperative pain and early quality of life after radiofrequency ablation and mechanochemical endovenous ablation of incompetent great saphenous veins. J Vasc Surg. 2013 Feb;57(2):445-50. doi: 10.1016/j.jvs.2012.07.049. Epub 2012 Nov 8. PMID 23141679
- [Result] Boersma D, van Eekeren RR, Werson DA, van der Waal RI, Reijnen MM, de Vries JP. Mechanochemical endovenous ablation of small saphenous vein insufficiency using the ClariVein((R)) device: one-year results of a prospective series. Eur J Vasc Endovasc Surg. 2013 Mar;45(3):299-303. doi: 10.1016/j.ejvs.2012.12.004. Epub 2013 Jan 9. PMID 23312507